CLINICAL TRIAL: NCT04458077
Title: Discover Learning - Social, Emotional and Identity Learning for Very Young Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Health for a Prosperous Nation (Other); Camara Education, Tanzania (Unknown); Ubongo Learning Limited (Unknown); Dalberg Global Development Advisors, Tanzania (Unknown); Save the Children (Other)
Responsible Party: Principal Investigator, Ronald Dahl, Director, Institute of Human Development, University of California, Berkeley
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-01-9464; OPP1158584 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Behavior, Adaptive; Behavior, Child; Behavior, Social
MeSH Terms: conditions — Behavior; Child Behavior; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile-phone-based SEIL Intervention (Experimental): This group will receive the Discover Learning 10-session intervention through a mobile-phone based platform over the course of 10 weeks (1 session per week).
  Interventions: Behavioral: Discover Learning (SEIL)

INTERVENTIONS:
Behavioral: Discover Learning (SEIL) — This mobile-phone-based intervention will assess the effectiveness of 10 SEIL sessions conducted at the household level with VYAs. Activities were designed to be done individually, with siblings/peers, and with parents/caregivers. This intervention will look at how household composition and types of practice that can enhance SEIL learning.

SUMMARY:
The primary aim of the Discover Learning Project (Discover) is to test an intervention for Very Young Adolescents (VYAs) to promote positive, gender norm transformative, social emotional and identity learning (SEIL). A secondary aim is to better identify effective components of Discover that are scalable requiring the lowest resources to implement

DETAILED DESCRIPTION:
This project builds on research from transdisciplinary developmental science that indicates that this period, which the investigators will call early adolescence (ages 10-14), is a period of dynamic maturational changes. These include the onset of pubertal development, which begins a period of rapid physical growth (including extensive brain development) and sexual maturation, as well as changes in cognitive, social, emotional, psychological, and behavioral processes. An emerging body of evidence supports the idea that this dynamic period of maturation is a sensitive period for social, emotional and motivational learning-in ways that can have enduring effects on a broad range of developmental trajectories including sexual and reproductive health, mental health, gender-based violence, education retention and attainment, and social development.

A foundational element of this research focuses on the social-emotional re-orientation of the developing brain at the onset of puberty, which appears to create natural affinities for discovery learning particularly in the social domain. In contrast to didactic learning models, discovery learning is a process through which learners engage in self-motivated inquiry, supported by teachers/facilitators, information and materials, in order to "discover" the intended content (Hammer, 1997). Key elements to creating sustainable discovery learning include: a) engaging motivation and natural curiosity and b) providing social scaffolding that includes a balance of monitoring/support while also promoting youth-driven discoveries (individually and in small groups). From a developmental science perspective, the beginning of puberty is associated with two important maturational changes that impact learning opportunities: 1) a general increase in the tendency to explore, discover, and to seek novelty/excitement; and 2) a particularly strong increase in natural curiosity to explore and understand one's larger social world, including social roles, social hierarchies, and an increased sensitivity to issues of social acceptance, admiration, and learning to establish key aspects of individual identity (Crone & Dahl, 2012). A core element to this early identity development is understanding oneself as a sexual and gendered individual in relation to those around her or him; accordingly, early learning experiences during this developmental window are fundamentally shaping the development of these identities in ways that have profound implications for all areas of health-especially sexual and reproductive health and vulnerability to gender-based exploitation and disadvantage.

The primary aim of this project is to develop and test the Discover Learning intervention with a goal of promoting positive, gender norm transformative, social-emotional learning during this crucial early window of opportunity. This work builds on developmentally informed principles that emphasize the importance of orchestrating a sensitive balance between promoting autonomy and providing adult engagement in ways that scaffold the discovery learning experience (Alifieri et al., 2011). The primary content (learning about interpersonal relationships and concepts of Social-Emotional Identity Learning) and method (introducing positive socially scaffolded exploration of the use of digital technology for youth-driven learning) have been chosen to strategically leverage this window of opportunity occurring during this sensitive period of learning. The approach is designed to help youth develop agency, become empowered, and to explore healthy pathways to finding meaning and purpose in their lives. To our knowledge, this is the first use of an integrative developmental science approach to leverage unique learning opportunities in early adolescence to impact broad improvements in health and education.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls currently enrolled in school/intervention site
* Ages 9-14

Exclusion Criteria:

* n/a

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Purpose from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from The Dimensions of Identity Development Scale (DIDS) (Mastrotheodoros & Motti-Stefanidi, 2017), validated self-reported instrument. Possible scores range from 0 (strongly disagree) to 3 (strongly agree) Change = Endline - Baseline score
Change in Emotional Self-Efficacy from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Adolescent Self Efficacy Questionnaire (Muris et.al, 2001), validated self-reported instrument. Possible scores range from 0 (not at all) to 4 (very well) Change = Endline - Baseline score
Change in Goal Orientation from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Goal Orientation Scale (Dowson and McInerney, 2004), validated self-reported instrument. Possible scores range from 0 (strongly disagree) to 4 (strongly agree) Change = Endline - Baseline score
Change in Persistence from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Persistence in Children (Lufi & Cohen, 1987), validated self-reported instrument. Possible scores range from 0 (strongly disagree) to 3 (strongly agree) Change = Endline - Baseline score
Change in Empathy from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Empathy (Overgaaw, et al, 2017), validated self-reported instrument. Possible scores range from 0 (not true) to 2 (often true) Change = Endline - Baseline score
Change in Internalizing Symptoms from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from African Youth Psychological Assessment (Betancourt, 2014), validated self-reported instrument. Possible scores range from 0 (never) to 3 (all the time) Change = Endline - Baseline score
Change in Externalizing Symptoms from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from African Youth Psychological Assessment (Betancourt, 2014), validated self-reported instrument. Possible scores range from 0 (never) to 3 (all the time) Change = Endline - Baseline score
Change in Academic Self-Efficacy from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Adolescent Self Efficacy Questionnaire (Muris et.al, 2001), validated self-reported instrument. Possible scores range from 0 (not at all) to 4 (very well) Change = Endline - Baseline score
Change in Curiosity from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Gender-free curiosity inventory (Reijo Byman, 2016), validated self-reported instrument in curiosity. Possible scores range from 0 (strongly disagree) to 3 (strongly agree) Change = Endline - Baseline score
Change in Teamwork from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Team Skills Index (Zhuang et al, 2008), validated self-reported instrument in curiosity. Possible scores range from 0 (never) to 3 (always) Change = Endline - Baseline score
Change in Growth Mindset from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Dweck's Theories of Intelligence (Growth Mindset Scale) (Ingebrigsten, 2018), validated self-reported instrument in curiosity. Possible scores range from 0 (never) to 3 (always) Change = Endline - Baseline score
Change in Outlook in Learning from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Dweck's Theories of Intelligence (Growth Mindset Scale) (Ingebrigsten, 2018), validated self-reported instrument in curiosity. Possible scores range from 0 (never) to 3 (always) Change = Endline - Baseline score
Change in Technology Perceptions from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Media and Technology Usage and Attitudes Scale (Rosen et al, 2013), validated self-reported instrument. Possible scores range from 0 (never) to 3 (always) Change = Endline - Baseline score
Change in Social Self-Efficacy from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Adolescent Self Efficacy Questionnaire (Muris et.al, 2001), validated self-reported instrument. Possible scores range from 0 (strongly disagree) to 3 (strongly agree) Change = Endline - Baseline score
Change in Prosocial Behavior from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from The Dimensions of Identity Development Scale (DIDS) (Mastrotheodoros & Motti-Stefanidi, 2017), validated self-reported instrument. Possible scores range from 1 (strongly disagree) to 4 (strongly agree) Change = Endline - Baseline score
Change in Gender Norms and Attitudes from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Discover Gender Norms and Attitudes Scale (under development), self-reported instrument. Possible scores range from 0 (strongly disagree) to 4 (strongly agree) Change = Endline - Baseline score
Change in Generosity from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Interpersonal Generosity Scale (IGS) (Smith & Hill, 2009), validated self-reported instrument. Possible scores range from 0 (strongly disagree) to 3 (strongly agree) Change = Endline - Baseline score
Change in Utu from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from Utu (under development), self-reported instrument. Possible scores range from 0 (strongly disagree) to 4 (strongly agree) Change = Endline - Baseline score
Change in Bullying from baseline to end of intervention | Baseline and endline, measured before the intervention and after the intervention (6 weeks)
  Standardized survey from The Global School-Based Students Health Survey (GSHS), validated self-reported instrument. Possible scores range from 0 (No) to 1 (Yes) Change = Endline - Baseline score

CONTACTS AND LOCATIONS:
Overall Officials: Ron Dahl, MD, Principal Investigator — Institute of Human Development
Locations (4):
- Tanzania (4):
  - Miburani Primary School, Dar es Salaam, Temeke
  - Sokoine Primary School, Dar es Salaam, Temeke
  - Twiga Primary School, Dar es Salaam, Temeke
  - Umoja Primary School, Dar es Salaam, Temeke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cherewick M, Lebu S, Su C, Richards L, Njau PF, Dahl RE. Study Protocol of a Distance Learning Intervention to Support Social Emotional Learning and Identity Development for Adolescents Using Interactive Mobile Technology. Front Public Health. 2021 Jan 28;9:623283. doi: 10.3389/fpubh.2021.623283. eCollection 2021. PMID 33585394
- [Derived] Cherewick M, Lebu S, Su C, Dahl RE. An Intervention to Enhance Social, Emotional, and Identity Learning for Very Young Adolescents and Support Gender Equity: Protocol for a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2020 Dec 31;9(12):e23071. doi: 10.2196/23071. PMID 33206624